CLINICAL TRIAL: NCT06663514
Title: SupporTive Care At Home Research : Single-center, Single-arm, Investigator-initiated Exploratory Clinical Trial for Patients with Neurologic Disease Patients
Brief Title: SupporTive Care At Home Research for Patients with Progressive Neurologic Disease Patients (STAHR-Neuro) (HOMECARE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BeLong Cho (Other)
Responsible Party: Sponsor-Investigator, BeLong Cho, professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HC21C0115-2
Record Dates: First submitted 2024-01-07; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-01

CONDITIONS: Supportive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: SupporTive Care At Home — Home-based medical care is based on a specialized home-based medical team approach, including following:
  Specialized Home-Based Medical Team Approach Initial Assessment and Education Initial Home Visits and Education Multidisciplinary Team Meeting Regular Assessment After the Initial Visit

SUMMARY:
To test the effects of home-based care on healthcare utilization within one Year (Hospitalization Status, Number of Hospitalizations, Unplanned Hospitalization Status, Number of Unplanned Hospitalizations, Length of Hospital Stay, Number of Emergency Room Visits, Number of Outpatient Visits) among progressive neurologic disease patients with decreased performance status. Home-based care includes education for patients and their family caregivers, home visits by specialized home-based medical staff, and regular status check-ups.

DETAILED DESCRIPTION:
This study is a Single-center, single-arm, investigator-initiated exploratory clinical trial to test the effects of home-based care on Healthcare Utilization within One Year (Hospitalization Status, Number of Hospitalizations, Unplanned Hospitalization Status, Number of Unplanned Hospitalizations, Length of Hospital Stay, Number of Emergency Room Visits, Number of Outpatient Visits)among neurologic disease Patients with decreased performance status. Home-based care includes education for patients and their family caregivers, home visits by specialized home-based medical staff, and regular status check-up. Study participants are recruiting from single institutions, aiming for 30 progressive neurologic disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Both the patient and their family caregiver must meet the criteria to be considered for this research.

Patient

Diagnosis of Progressive Neurological Disorders (Motor Neuron Disease, Parkinson's Disease) with ICD-10 codes (G12.2, G20, G11.9, G21, G22, G23, G30.8, G31.8, F02.3, etc.), additional diseases can be included depending on the patient's condition.

Individuals with a modified Rankin Score (mRS) of 3-5 A person who wishes to stay at home A person whose family caregiver resides at home A person who wishes to participate in the research Family Caregiver

A family* member of the patient

* Family: refers to the patient's spouse (including a common-law partner), descendants and their spouses up to the second degree, siblings and their spouses, and relatives and their spouses up to the eighth degree.

A person who meets one of the following conditions:

Lives with the patient (patient's household member) Does not live with the patient, but visits the patient's home more than three times a week A person who wants the patient to stay at home A person who can communicate easily with medical staff A person who wishes to participate in the research

Exclusion Criteria:

* If either the patient or the family caregiver meets any one of these criteria, they are excluded from the study.

Patient

A person who cannot speak, hear, or read Korean A person who is judged by a medical doctor to be unable to take part in this research due to extremely poor health A person residing outside the range that can be visited by the respective medical institution (the conditions for distance are to be specified by each medical institution)*

* This condition is not applicable for the control group.

A person who has used hospital- or home-type hospice and palliative care services A person who is under the age of 19 Family Caregiver

A person who cannot speak, hear, or read Korean A person who is judged by a medical doctor to be unable to take part in this research due to extremely poor health A person under the age of 19

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Unplanned hospitalization | within One Year
  admission to the enrolled hospital to treat unexpected symptoms or medical conditions (not including planned admission for chemotherapy or admission for planned surgery or intervention) admission to a hospital other than the enrolled hospital admission to a nursing hospital for a duration of less than 4 weeks.

SECONDARY OUTCOMES:
Patient medical utilization | within 12 months following enrollment
  The total number of hospital utilization, including hospitalization, emergency room visit, and clinic visits
Hospitalization | within 12 months following enrollment
  the number of hospitalization
ER visits | within 12 months following enrollment
  the number of emergency room visits
Healthcare use | within 12 months following enrollment
  the number of healthcare use for severe diseases
Patient end-of-life care: ICU admission | within 1 month before death
  ICU admission one month before death
Patient end-of-life care: ventilator treatment | within 1 month before death
  Mechanical ventilator apply one month before death
Patient end-of-life care: an advance directive | within 1 month before death
  Completion of advance medical directives within 1 month before death
symptom management | within 12 months following enrollment
  IPOS-neuro S8 of patient
Quality of life of patient - EQ-5D | within 12 months following enrollment
  Euro-Quality of Life-5 Dimension (EQ-5D) of patient
Satisfaction with services (patient) | within 12 months following enrollment
  Satisfaction of the study participant (patient) with the service in this study, evaluated by questionnaire
Quality of life of family caregiver | within 12 months following enrollment
  Euro-Quality of Life-5 Dimension (EQ-5D) of family caregiver
Care burden of family caregiver | within 12 months following enrollment
  The Korean version of Caregiver Reaction Assessment (CRA-K) of family caregiver
Depressive symptom of family caregiver | within 12 months following enrollment
  Patient Health Questionnaire-9 (PHQ-9) of family caregiver
Caring competency of family caregiver | within 12 months following enrollment
  Caring competency of family caregiver, measured by questionnaire
Satisfaction with services (family caregiver) | within 12 months following enrollment
  Satisfaction of the study participant (family caregiver) with the service in this study, evaluated by questionnaire
Expenses | within 12 months following enrollment
  medical expenses, care expenses

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No